CLINICAL TRIAL: NCT03671538
Title: A Randomized Phase II Study of Anlotinib Combined With Pemetrexed and Cisplatin in First Treatment for Advanced Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor Negative Mutations
Brief Title: Non Squamous NSCLC Patients With Anlotinib Combined With Pemetrexed and Cisplatin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lingyu Luo (Other)
Responsible Party: Sponsor-Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L008
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — anlotinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Plus Pemetrexed and Cisplatin (Experimental): pemetrexed 500mg/m2 and Cisplatin 75mg/m2 on day 1 of a 21-day cycle ;Anlotinib 12mg qd on day 1 to 14 of a 21-day cycle
  Interventions: Drug: Anlotinib; Drug: pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 12mg qd on day 1 to 14 of a 21-day cycle
Drug: pemetrexed — pemetrexed 500mg/m2 on day 1 of a 21-day cycle ;
Drug: Cisplatin — Cisplatin 75mg/m2 on day 1 of a 21-day cycle ;

SUMMARY:
Chemotherapy is still the standard first-line treatment option for EGFR unmutated patients. After a randomized phase Ⅲ trial, BEYOND was presented the synergistic effect of progression-free survival(PFS) could be expected when chemotherapy is combined with Antiangiogenesis agent bevacizumab in China;Therefore,in this study, The investigators will investigate the efficacy and safety of Anlotinb combined With Pemetrexed and Cisplatin as first-line therapy in patients with chemotherapy-naive, stage IIIB or IV, non-squamous NSCLC without targetable EGFR or ALK genetic aberrations.

DETAILED DESCRIPTION:
This is a randomized, single -center study conducted in China to compare the efficacy and safety of Anlotinb combined With Pemetrexed and Cisplatin as first-line therapy in patients of Advanced Gene Negative Non-squamous Non-small Cell Lung Cancer.

Eligible patients will be randomized to arm A:

Patients were instructed to take 500mg/m2 pemetrexed as a 10-minute intravenous infusion and Cisplatin 75mg/m2 on day 1 of a 21-day cycle and12mg Anlotinib orally daily on day 1 to 14 of a 21-day cycle.If there was no evidence of disease progression following a maximum of 4-6 cycles of anlotinib plus chemotherapy, patients continued to receive single-agent anlotinib until disease progression or unacceptable toxicity. Approximately 62 patients will be enrolled to ensure complete treatments for primary endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

* Be≥18 years of age on the day of signing informed consent and With good compliance and agree to accept follow-up of disease progression and adverse events.
* Patients with histologic or cytologic confirmation of advanced or metastatic Non squamous NSCLC with stage IIIB or IV disease.（For recurrent patients, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment）
* Patients have not been received systematic treatment，including chemotherapy and EGFR-TKIs
* EGFR mutations confirmed by molecular detection (including, but not limited to, T790M, 19 exon deletion and L858R) external pathological examination was accepted (including pathological or blood test results)
* There were at least one target lesions in the past three months has not yet accepted radiotherapy, and could be recorded by magnetic resonance imaging (MRI) or computer tomography (CT) measuring accurately at least in one direction(The maximum diameter needs to be recorded), including conventional CT ≥20 mm or spiral CT ≥10 mm.
* Life expectancy ≥3 months.
* Have a performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* With normal marrow, liver ,renal and coagulation function:
* The blood routine examination need to be standard (no blood transfusion and blood products within 14 days, no g-csf and other hematopoietic stimulating factor correction)
* Hemoglobin（HB）≥90 g/L
* A Neutrophil count of （ANC）≥1.5×109/L
* A Platelet count of （PLT）≥80×109/L
* A total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL)
* A alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL, in case of liver metastasis ALAT and ASAT≤5 UNL
* A creatinine (Cr) of ≤1.5 UNL; a creatinine clearance rate ≥ 60ml/min (Cockcroft-Gault)
* Doppler echocardiography: left ventricular ejection fraction (LVEF) is lower than normal (50%)
* Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug.

Exclusion Criteria:

* Small cell lung cancer (include Small cell lung cancer mixture of NSCLC)
* Iconography (CT or MRI) shows that the tumor vessels have 5 mm or less, or Cardiovascular involvement by Central tumor ; Or obvious lung empty or necrotic tumor
* Patients with Other active malignant tumors requiring concurrent treatment;
* Patients has a history of malignant tumors. Patients with basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma, or cervical cancer in situ who have undergone possible curative treatment and have not suffered any recurrence of the disease within 5 years from the start of treatment
* Patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination revealed brain or leptomeningeal disease） (14 days before the random treatment has been completed and the symptoms of patients with brain metastases from stable can into the group, but need to the cerebral MRI, CT or vein angiography confirmed as without symptoms of cerebral hemorrhage).
* Patients who have not recovered to grade 1 or below according to NCI-CTCAE4.0 after previous systemic antitumor therapy (except alopecia)
* Uncontrollable hypertensive (systolic blood pressure or greater 140 mmHg or diastolic blood pressure or greater 90 mmHg, despite the best drug treatment)
* Patients with NCI-CTCAE grade II or greater peripheral neuropathy, except due to trauma
* Significant cardiac disease as defined as: grade II or greater myocardial infarction, unstable arrhythmia(Including corrected QT interval (QTc )period between male or greater 450 ms, female or greater 470 ms); New York Heart Association (NYHA) grade II or greater heart dysfunction , or Echocardiography reveal left ventricular ejection fraction （LVEF）Less than 50%
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or be treated with thrombolysis and anticoagulation. Note: under the premise of International Normalized ratio (INR) of prothrombin time (PT) Less than or equal to 1.5, allow to administrate low-dose heparin (adult daily dose is 06000 ~ 12000 U) or low-dose aspirin (100 mg daily dosage or less) , for prophylactic purposes.
* Urine routines show urine protein≥ ++, or urine protein quantity≥ 1.0 g during 24 hours
* Patients with severe infections , and need to receive systemic antibiotic treatment.（according to the CTC AE4.0, the infection with grade 2 or above and requiring intravenous antibacterial therapy ）;Decompensated diabetes or other contraindication with high dose glucocorticoid therapy）
* Patients with respiratory syndrome (difficulty breathing of level 2 or higher according to the CTC AE), serous cavity effusion need to surgical treatment (according to the CTC AE4.0, including pleural of level 2 or higher with respiratory distress and anoxia, need for intubation or pleurodesis treatment, severe ascites of level 2 need to surgery invasive treatment, pericardial of level 2 and affect physiological function)
* Serious, non-healing wound, ulcer, or bone fracture
* Active or chronic hepatitis c and/or Hepatitis B virus (HBV) infection
* Has an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* Has received major surgery or severe traumatic injury, fractures or ulcer Within 4weeks before Random
* Patients have participated in other antitumor drug clinical trials Within 4 weeks before enrollment or prepare to receive systemic anti-tumor treatment during the study or Within 4 weeks before randomization, including cytotoxic therapy cellular, Signal transduction inhibitors, immune therapy (or receiving mitomycin C Within six weeks before taking experimental drug therapy).Field overspread radiotherapy (ef-rt) was carried out within 4 weeks before the grouping or limited field radiotherapy was carried out within 2 weeks before the grouping to evaluate tumor lesions
* Severe weight loss (> 10%) Within 6 weeks before Random
* Has Clinically significant hemoptysis Within 3 months before Random (daily hemoptysis than 50 ml;Or significant clinical significance of bleeding symptoms or have definite bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers, baseline period + + and above of fecal occult blood, or vasculitis, etc
* Has venous thromboembolism events Within 12 months before Random, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | From enrollment to completion of study. Estimated about 24 months.
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Overall Response Rate | From enrollment to progression of disease. Estimated about 24 months
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, Overall Response Rate)
disease control rate | From enrollment to progression of disease. Estimated about 24 months
  Clinical response of treatment according to RESIST v1.1 criteria (DCR, disease control rate)
Overall Survival | From enrollment to completion of study. Estimated about 24 months.
  From date of randomization until the date of death or date of last visit/contact, whichever came first
6-month PFS rate | From enrollment to analysis, Estimated about 6 months
  Proportion of people who first documented disease progression or death from any cause, whichever came first ,during 6 months
12-month PFS rate | From enrollment to analysis. Estimated about 12 months.
  Proportion of people who first documented disease progression or death from any cause, whichever came first ,during 12 months